CLINICAL TRIAL: NCT03802864
Title: Post-operative Pain Control of Testicular Sperm Extraction Using Liposomal Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1802018993
Record Dates: First submitted 2019-01-04; First posted 2019-01-14 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: The study model is a randomized double blind control trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine (Experimental): Participants in this arm will have a single injection of liposomal bupivacaine admixed with standard bupivacaine (266mg liposomal bupivacaine mixed with 50mg bupivacaine hydrochloride) at the conclusion of their surgical sperm retrieval procedure.
  Interventions: Drug: Liposomal Bupivacaine
- Standard Bupivacaine (Active Comparator): Participants in this arm will have a single injection of standard bupivacaine (100mg bupivacaine hydrochloride) at the conclusion of their surgical sperm retrieval procedure.
  Interventions: Drug: Standard Bupivacaine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — After surgical sperm retrieval, the wound will be injected with liposomal bupivacaine (266 mg) mixed with standard bupivacaine (bupivacaine hydrochloride 50mg) for post-operative pain relief.
  Arms: Liposomal Bupivacaine
Drug: Standard Bupivacaine — After surgical sperm retrieval, the wound will be injected only with standard bupivacaine (bupivacaine hydrochloride 100mg) for post-operative pain relief.
  Arms: Standard Bupivacaine

SUMMARY:
The study is a drug trial comparing the post-operative pain control provided by liposomal bupivacaine (a local anesthetic) against standard bupivacaine (a different formulation of the local anesthetic) for men undergoing testicular sperm extraction.

ELIGIBILITY:
Inclusion Criteria:

* Men scheduled for surgical sperm retrieval for infertility
* Men 18 years and older who can provide informed consent
* No documented allergy to bupivacaine or celecoxib

Exclusion Criteria:

* Prior history of substance abuse
* Any narcotic use within the last 3 months
* Concomitant use of aspirin
* Any of the following comorbidities: renal failure, heart disease, peptic ulcer disease, cerebrovascular disease, significant liver disease, untreated depression, chronic pain disorder, or bleeding diatheses
* Medical history or concurrent illness that the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial, or constitutes an unacceptable risk to the subject

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Hayden, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine Department of Urology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (9.3) | 36.4 (11.9) | 36.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 22 | 19 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores 48 Hours After Surgery
Description: Every 8 hours in the first 48 hours post-surgery, subjects were prompted to report their pain score on the 11-point numerical pain rating scale, NRS-11 (Numerical Rating Scale, 11 points). 0 indicates no pain and 10 indicates worst possible pain.
  Each subject's pain scores were then plotted against time, and the area under the curve was then computed. The minimum composite score would be 0 (no pain ever reported), and the maximum composite score would be 480 (maximum pain (score of 10) reported each time across 48 hours).
Time Frame: First 48 hours after surgery
Measure: Mean (Standard Deviation); unit: Scores*Hour
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 25 | 25
Scores*Hour | 118.4 (99.7) | 98.2 (68.9)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Superiority; p = 0.41, t-test, 2 sided

2. Secondary Outcome: Pain Scores 60 Hours After Surgery
Description: Every 12 hours in the first 60 hours post-surgery, subjects were prompted to report their pain score on the 11-point numerical pain rating scale, NRS-11 (Numerical Rating Scale, 11 points). 0 indicates no pain and 10 indicates worst possible pain.
  Each subject's pain scores were then plotted against time, and the area under the curve was then computed. The minimum composite score would be 0 (no pain ever reported), and the maximum composite score would be 600 (maximum pain (score of 10) reported each time across 60 hours).
Time Frame: First 60 hours after surgery
Measure: Mean (Standard Deviation); unit: Scores*Hour
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 25 | 25
Scores*Hour | 140.7 (107.8) | 116 (83.2)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Superiority; p = 0.37, t-test, 2 sided

3. Secondary Outcome: Pain Scores 7 Days After Surgery
Description: Every 12 hours in the first 7 days post-surgery, subjects were prompted to report their pain score on the 11-point numerical pain rating scale, NRS-11 (Numerical Rating Scale, 11 points). 0 indicates no pain and 10 indicates worst possible pain.
  Each subject's pain scores were then plotted against time, and the area under the curve was then computed. The minimum composite score would be 0 (no pain ever reported), and the maximum composite score would be 1680 (maximum pain (score of 10) reported each time across 168 hours).
Time Frame: First 7 days after surgery
Measure: Mean (Standard Deviation); unit: Scores*Hour
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 25 | 25
Scores*Hour | 286.6 (202.7) | 233.1 (209.9)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Superiority; p = 0.36, t-test, 2 sided

4. Secondary Outcome: Narcotic Requirement
Description: Total number of narcotic tablets required between the intervention and control arms during post-operative day 1 through 7.
Time Frame: First 7 days after surgery
Measure: Mean (Standard Deviation); unit: Count of narcotic tablets
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 25 | 25
Count of narcotic tablets | 2.6 (4.4) | 1.6 (3.1)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Superiority; p = 0.28, Regression, Linear

5. Secondary Outcome: Time to Narcotic Rescue
Description: Time (in hours) to first rescue narcotic utilization between the two arms.
Time Frame: First 7 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 25 | 25
Participants
  0 to 40 Hours After Surgery | 10 | 8
  41 to 80 Hours After Surgery | 0 | 0
  81 to 120 Hours After Surgery | 0 | 3
  121 to 160 Hours After Surgery | 2 | 1
  Never Required Narcotics | 13 | 13
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Superiority; p = 0.78, Log Rank

6. Secondary Outcome: Pain Control Satisfaction
Description: Overall satisfaction of pain control regimen self reported on post-operative day 7. The prompt required a yes/no answer. The percent of participants answering "yes" will be compared between the two arms.
Time Frame: 7th day after surgery
Population: 3 subjects from the Liposomal Bupivacaine arm and 4 subjects from the Standard Bupivacaine arm weren't analyzed because they didn't provide answers to the yes/no prompt.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 22 | 21
Participants
  Yes - Adequate pain control achieved | 22 | 20
  No - Adequate pain control not achieved | 0 | 1
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Superiority; p = 0.49, Fisher Exact

7. Secondary Outcome: Percentage of Patients Not Requiring Any Narcotics
Description: The percentage of patients remaining opiate free by post-operative day 7.
Time Frame: 7th day after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 25 | 25
Participants
  No narcotics required | 15 | 16
  Narcotics required | 10 | 9
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Superiority; p = 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events from the time of their initial surgery until 3 weeks after surgery.
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/25 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine (N=25) | Standard Bupivacaine (N=25)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Scrotal Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal infection (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT03802864/Prot_SAP_000.pdf